CLINICAL TRIAL: NCT05310448
Title: Tumor Treating Fields: Pilot Study of Adjuvant Treatment for Brainstem Gliomas
Brief Title: Tumor Treating Fields for the Treatment of Brainstem Gliomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jim Zhong, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003027; NCI-2021-09679 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP5412-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-02-04; First posted 2022-04-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (tumor treating fields) (Experimental): After completion of standard of care radiation therapy, patients wear the Optune device for 18 hours per day for 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Device: Optune device

INTERVENTIONS:
Device: Optune device — Wear Optune device
  Other Names: Alternating Electric Field Therapy; TTF; TTFields; Tumor Treating Fields Therapy

SUMMARY:
This clinical trial tests the safety and side effects of tumor treating fields in treating patients with gliomas located in the brainstem. Optune is a wearable, portable, treatment that creates low-intensity, wave-like electric fields called tumor treating fields (TTFields), which interfere with cancer cell division. TTFields may prevent growth or decrease size of gliomas in patients

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of tumor treating fields in combination with standard of care radiotherapy and chemotherapy in patients with brainstem gliomas.

SECONDARY OBJECTIVE:

I. To evaluate the anti-tumor activity of the combination of radiotherapy, chemotherapy, and tumor treating fields by assessing progression-free survival (PFS), overall response rate, and overall survival (OS).

TERTIARY/EXPLORATORY OBJECTIVE:

I. To assess the effects of the tumor treating fields on neurocognitive function.

OUTLINE:

Beginning after start of standard of care radiation therapy, patients wear the Optune device for at least 18 hours per day for 12 months in the absence of disease progression or unacceptable toxicity.

During study treatment, patients are followed up at 3, 6, 9, and 12 months. After study treatment, patients are followed up every 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Karnofsky performance status >= 70%
* Life expectancy > 12 weeks as determined by the investigator
* Diagnosis of glioma with at least partial involvement or invasion of thalamus, cerebral peduncles, midbrain, pons, or medulla. Confirmation of diagnosis by biopsy or maximal safe resection preferred. If multi-disciplinary tumor board recommend no benefit and likely harm of attempting biopsy then can establish consensus clinical diagnosis. If foregoing biopsy then tumor board will estimate tumor stage based on clinical presentation and radiographic findings.
* Completion of all previous therapy (including surgery and radiotherapy) for the treatment of cancer >= 4 weeks before the start of study therapy.
* Willingness and ability of the subject to comply with scheduled visits, drug administration plan, protocolspecified laboratory tests, other study procedures, and study restrictions.
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation.
* Patients must have adequate organ and marrow function, within 28 days of Cycle 1 Day 1 of Temozolomide, as defined below:

Hematology:

* Hemoglobin >= 9.0 g/dl (no transfusions allowed within 7 days of cycle 1 day 1 to meet entry criteria) (within 28 days of cycle 1 day 1 of temozolomide)
* White blood cell (WBC) >= 2000/uL (after at least 7 days without growth factor support or transfusion) (within 28 days of cycle 1 day 1 of temozolomide)
* Absolute neutrophil count (ANC) >= 1,500/mcL (after at least 7 days without growth factor support or transfusion) (within 28 days of cycle 1 day 1 of temozolomide)
* Platelets >= 100,000/mcL (no transfusions allowed within 7 days of cycle 1 day 1 to meet entry criteria) (within 28 days of cycle 1 day 1 of temozolomide)
* Prothrombin time (PT)/partial thromboplastin time (PTT) =< 1.5 x upper limit of normal (ULN) (within 28 days of cycle 1 day 1 of temozolomide)

Chemistry

* Total bilirubin =< 2 institutional upper limit of normal (ULN) (within 28 days of cycle 1 day 1 of temozolomide)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 institutional upper limit of normal (ULN) (within 28 days of cycle 1 day 1 of temozolomide)
* Serum creatinine =< 2 mg/dL (or glomerular filtration rate >= 40 mL/min) (within 28 days of cycle 1 day 1 of temozolomide)
* The effects of combination therapy with tumor treating fields (TTF) and temozolomide on the developing human fetus are unknown. For this reason and because other therapies used in this trial are known to be teratogenic, female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy.
* FCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 12 months after completion of TTF and Temozolomide administration. A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

- Patients who have completed chemotherapy or radiotherapy more than 26 weeks prior to entering the study.

i. Completion of radiotherapy 8-12 weeks prior to starting the tumor treating fields will be considered a minor deviation.

ii. Completion of radiotherapy 13-26 weeks prior to starting the tumor treating fields will be considered a major deviation.

* Patients who are receiving any other investigational agents or an investigational device within 21 days before first administration of study device.
* History of allergic reactions attributed to compounds of similar composition to those used for transducer placement.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Significant cardiovascular disease (eg, myocardial infarction, arterial thromboembolism, cerebrovascular thromboembolism) within 3 months prior to start of study therapy; angina requiring therapy; symptomatic peripheral vascular disease; New York Heart Association Class 3 or 4 congestive heart failure; or uncontrolled Grade ≥3 hypertension (diastolic blood pressure ≥100 mmHg or systolic blood pressure ≥160 mmHg) despite antihypertensive therapy.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of increased risk of lethal infections when treated with marrow-suppressive therapy such as Temozolomide. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 12 months after TTFields started
  Adverse event rates will be summarized descriptively using frequencies and percentages in addition to a tolerability rate defined as composite of any dose-limiting toxicity.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From TTFields start to disease progression or death, assessed up to 36 months
  PFS will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median PFS will be estimated using the Brookmeyer-Crowley approach.
Overall response rate | Up to 12 months after TTFields started
  Evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Overall survival (OS) | From TTFields start to death from any cause, assessed up to 36 months
  OS will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median OS will be estimated using the Brookmeyer-Crowley approach.

CONTACTS AND LOCATIONS:
Overall Officials: Jim Zhong, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (3):
- United States (3):
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia